CLINICAL TRIAL: NCT03685266
Title: Efficiency of Task Switching and Multi-tasking: Observations of Pediatric Resident Behaviors When Managing Interruptions to Daily Workflow
Brief Title: Efficiency of Task Switching and Multi-tasking
Status: Completed | Type: Observational
Sponsor: University of Hawaii (Other)
Responsible Party: Principal Investigator, Jennifer Di Rocco, Assistant Professor, University of Hawaii
Other Study IDs: 2015-107
Record Dates: First submitted 2016-05-17; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Task Performance and Analysis; Efficiency
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Residents: Participating pediatric residents from first postgraduate year (PGY-1) through third postgraduate year (PGY-3) will be observed over a 12 month timeframe.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — There are no specific interventions in this study; it is observational only. One could argue that the act of observing the participants may change their behavior (the Hawthorne effect).

SUMMARY:
This study will collect observational data on how well pediatric residents handle interruptions to their daily workflow. Residents will be directly observed during their work day and behaviors will be recorded using an electronic tool that will time-stamp their actions when faced with an interruption. The average time it takes for them to return to their original task(s) after faced with an interruption will be calculated, along with correlations made between their predicted multi-tasking ability, year of training, and additional factors.

DETAILED DESCRIPTION:
Efficiency of Task Switching and Multi-tasking: Observations of Pediatric Resident Behaviors when Managing Interruptions to Daily Workflow

Jennifer R. Di Rocco, DO, Assistant Professor of Pediatrics, JABSOM; Associate Program Director, UH Pediatric Residency Program; Master of Education Candidate, University of Cincinnati/Cincinnati Children's Hospital

Summary of Project Concept:

The daily practice of medicine is fraught with frequent interruptions that a busy clinician must manage appropriately in order to ensure the best patient care possible. Tasks that are urgent and time-sensitive must be prioritized, organized, and balanced with numerous other tasks requiring completion during the day. Physicians must also maintain the necessary flexibility required to adapt to unexpected events that inevitably surface regularly during a busy clinical workday. The ability to expertly manage interruptions may be considered under the umbrella of the "art of medicine," which is not found in textbooks and can be difficult to teach. Additional challenges in this era of limited duty hours include limited patient exposure with less time to develop the skills for effective management of interruptions. Some young clinicians seem to easily triage tasks as they are presented, while others struggle with this role.

Pediatric residents have graded autonomy as they progress through a program, with a steep learning curve in their first year. From an initial dependence on the senior resident and faculty when starting as a new intern to improved ability to independently practice as they near the start of their second year, each intern matures both clinically and professionally at various rates. The Accreditation Council of Graduate Medical Education (ACGME) has assigned 21 pediatric milestones that must be reported back to them twice yearly with a resident's progress along the continuum. Milestones describing the degree of medical knowledge, trustworthiness, leadership, teamwork and stress management skills are all required and applicable to the topic of one's ability to manage interruptions appropriately. The description of the "Patient Care 2" milestone, which reads "Organize and prioritize responsibilities to provide patient care that is safe, effective and efficient" addresses the concept of the "optimization of multitasking" in the milestone discussion. This is described as a higher level of clinical achievement in which a physician demonstrates concurrent task completion in a manner ends to a more efficient workflow without compromising patient safety. The complex set of behaviors described by this milestone can be best observed and assessed when a resident has increased responsibility and leadership roles including supervising a team, managing pager calls and admitting new patients simultaneously. Some residents in our program in recent years have struggled in supervisory roles, specifically with this milestone, but some have excelled, despite having less practice than prior decades of trainees. Understanding the factors contributing to how pediatric residents manage interruptions (from "novice" interns to "expert" third year residents) should be helpful towards designing curricula for mastery of these skills in our program and in others across the nation.

Many factors are involved in how physicians manage interruptions, and the positive or negative effects of their management decisions have implications on patient safety and medical errors in the clinical workplace. Observational studies of pediatric residents do not exist in the current literature, nor does a study exist that correlates physicians' ability and quality of interruption management with their overall wellness including their preferred learning styles, aptitudes in dealing with interruptions, sleep debt, and mental strain. Garnering such data and analyzing such variables could provide added guidance and understanding to those residency programs that are struggling to help learners improve in this arena, which is difficult to truly assess until a resident is in a supervisory position with multifactorial responsibilities. If there were a way of predicting aptitude in this skill set early, learners who may not easily manage interruptions could be targeted and practice exercises designed to strengthen this skill set. With this intervention, the transition from an intern to a senior supervising resident may be much smoother. The first step towards creating tools for augmenting performance in the area of managing interruptions gracefully and efficiently is to understand the current factors that are involved in a resident's decision process when faced with interruptions during the daily workflow. An observational study of residents in real time would provide such data and serve as a springboard for future work in creating tools and curricula to assist residents struggling with task management.

Project methods will include IRB approval and recruitment of pediatric residents. Participants will be asked to complete some baseline surveys (which include wellness and sleep inventories) and a multitasking exercise (called the Multitasking Assessment Tool or MTAT). Residents will then be observed multiple times over 1-2 hour time slots when rotating in both the general pediatric wards and emergency department settings by the study leader or by a trained observer, with all behaviors categorized and recorded with time stamps via a portable electronic database time-motion tool. On the day of observation, each participant will complete two short surveys regarding the degree of stress they are feeling that day as well as a log of their previous week's sleep habits.

ELIGIBILITY:
Inclusion Criteria:

* Consenting pediatric residents

Exclusion Criteria:

* Non-consenting pediatric residents

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All pediatric residents at the University of Hawai'i Pediatric Residency Program will be recruited as potential participants.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
MTAT score predicting residents who take the least time to return to an original task after an interrupting task | Through study completion, up to 1 year
  Hypothesis: A lower, more efficient MTAT score will predict the most efficient residents, as defined by taking the least amount of time to manage interruptions as directly observed and recorded through a time-motion tool.

SECONDARY OUTCOMES:
Time to return to task after interruption | Through study completion, up to 1 year
  Hypothesis: Senior level pediatric residents will take less time to return to an original task following an interrupting task as compared to first year residents.
Self-assigned level of personal wellness affects task-switching efficiency | Through study completion, up to 1 year
  Hypothesis: Yes, low wellness scores, as individually self-reported on a scale of 0-10 negatively impact task-switching efficiency.

OTHER OUTCOMES:
Self-reported hours of sleep affects task-switching efficiency | Through study completion, up to 1 year
  Hypothesis: Yes, lower average hours of sleep, as individually self-reported in hours of sleep each day in the preceding week, negatively impact task-switching efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Di Rocco, DO, Principal Investigator — University of Hawai'i
Locations (1):
- Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carraccio C, Benson B, Burke A, Englander R, Guralnick S, Hicks P, Ludwig S, Schumacher D, Vasilias J. Pediatrics milestones. J Grad Med Educ. 2013 Mar;5(1 Suppl 1):59-73. doi: 10.4300/JGME-05-01s1-06. No abstract available. PMID 24404214
- See also: Background and information about the Multitasking Assessment Tool (MTAT) — http://www.multitaskingtests.com